CLINICAL TRIAL: NCT05562791
Title: Pilot Study of 68Gallium PSMA-PET/CT in Patients With Metastatic Urothelial Carcinoma or Melanoma
Brief Title: A Study of 68Gallium PSMA-PET/CT Scans in People With Bladder Cancer or Skin Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-157
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
Keywords: Metastatic; Urothelial carcinoma; 68Gallium; PSMA-PET/CT; 22-157
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis; Carcinoma, Transitional Cell | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm pilot study of 68Gallium PSMA-PET/CT imaging in patients with metastatic urothelial carcinoma or Melanoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with metastatic urothelial carcinoma lesions (Experimental): Patients will initially undergo a standard of care FDG PET with diagnostic CT scan followed by an investigational 68Ga PSMA PET/CT scan.
  Interventions: Drug: [68Ga]PSMA; Diagnostic Test: PET/CT imaging
- Patients with melanoma lesions (Experimental): Patients with melanoma who have 1 or more radiographically assessable metastatic lesions on standard of care imaging will undergo a 68Gallium PSMA-PET/CT and standard of care imaging (either FDG PET or CT scan).
  Interventions: Drug: [68Ga]PSMA; Diagnostic Test: PET/CT imaging

INTERVENTIONS:
Drug: [68Ga]PSMA — 68Gallium PSMA-PET/CT imaging within 10 days after standard of care FDG-PET/CT.
Diagnostic Test: PET/CT imaging — 68Gallium PSMA-PET/CT imaging within 10 days after standard of care FDG-PET/CT.

SUMMARY:
The purpose of this study is to see whether 68Gallium PSMA-PET/CT scans are an effective way to detect sites of cancer in people with metastatic bladder cancer or skin cancer. The study researchers want to learn if a 68Gallium PSMA PET/CT scan will work better, the same, or not as well as the PET/CT scans doctors usually use for imaging bladder cancer or skin cancer (FDG-PET/CT scan).

ELIGIBILITY:
Inclusion Criteria for Urothelial Carcinoma Cohort:

* Patients with histologically confirmed metastatic urothelial carcinoma with extrapelvic nodal and/or visceral sites of disease (including lung, liver, bone, or soft tissue)
* At least 3 lesions assessable by FDG PET/CT according to RECIST and PERCIST guidelines where applicable, that are determined suspicious for metastasis by an MSKCC attending radiologist or nuclear medicine physician.
* Karnofsky performance status ≥50% (or ECOG/WHO ≤2)
* Participant is ≥18 years of age
* Patient must be able to understand and is willing to sign a written informed consent document

Inclusion Criteria for Melanoma Cohort:

* Patients with histologically confirmed metastatic melanoma
* At least 1 metastatic lesion assessable by CT or FDG PET/CT according to RECIST that is determined to be suspicious for metastasis by an MSKCC attending radiologist or nuclear medicine physician
* ECOG <= 2
* Participant is >= 18 years of age
* Patient must be able to understand and is willing to sign a written informed consent document

Exclusion Criteria for Urothelial Carcinoma Cohort:

* Patients with pelvic node-only metastatic disease. If the patient has lymph node only disease, at least one PET-assessable node must be located outside of the pelvis
* Patients with bone only disease
* Unable to lie flat, still, or to tolerate a PET scan
* Patient undergoing active treatment for non-urothelial malignancy, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized.
* Patients on a therapeutic clinical trial where PSMA imaging would interfere with the conduct of the trial
* Patients undergoing active surveillance with a known history of non-urothelial malignancies
* Women who are pregnant. All women of childbearing potential must have a documented negative pregnancy test.

Exclusion Criteria for Melanoma Cohort:

* Unable to lie flat, still, or tolerate PET scan.
* Patient is on another therapeutic trial where PSMA imaging would interfere with the conduct of the trial.
* Women who are pregnant. All women of childbearing potential must have a documented negative pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Define the proportion of patients with 1 or more lesions detectable by 68Gallium PSMA-PET/CT for Urothelial Carcinoma | 1 year
  If 6 of 10 patients have at least one lesion identified both on standard of care FDG PET/CT and also detected on 68Gallium PSMA-PET/CT, this imaging modality will be worthy of further exploration in metastatic UC.
Define the proportion of patients with 1 or more lesions detectable by 68Gallium PSMA-PET/CT for Melanoma | 1 year
  If 6 of 10 patients have at least one lesion identified both on standard of care FDG PET/CT and also detected on 68Gallium PSMA-PET/CT, this imaging modality will be worthy of further exploration in metastatic Melanoma.

CONTACTS AND LOCATIONS:
Overall Officials: Gopakumar Iyer, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm